CLINICAL TRIAL: NCT06469268
Title: Development and Application Study of ePRO (Patient Reported Outcome) Software for Managing Cancer Patients Throughout the Treatment Period
Brief Title: Development and Application Study of ePRO Software for Managing Cancer Patients Throughout the Treatment Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shikai Wu (Other)
Responsible Party: Sponsor-Investigator, Shikai Wu, Director of Oncology Department, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ePRO-001
Record Dates: First submitted 2024-05-29; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult
Keywords: Epro; peritherapeutic period; safety; Efficacy

STUDY DESIGN:
Intervention Model Description: Enrolled patients who received cisplatin or oxaliplatin were randomly assigned to one of two groups. Group A was the routine observation group, 50 patients were enrolled in the group. After receiving antineoplastic drug treatment, they were discharged home, and the treatment-related adverse reactions were observed and intervention according to the routine process. Group B was the ePRO study group: A total of 50 patients were enrolled in this group. After receiving anti-tumor drug treatment, the ePRO system was installed through the mobile phone. After training, the patients could skillfully use the ePRO system.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): This was the routine observation group, 50 patients were enrolled in the group. After receiving antineoplastic drug treatment, they were discharged home, and the treatment-related adverse reactions were observed and intervention according to the routine process.
- Group B (Experimental): This was the ePRO study group: A total of 50 patients were enrolled in this group. After receiving anti-tumor drug treatment, the ePRO system was installed through the mobile phone. After training, the patients could skillfully use the ePRO system.
  Interventions: Device: Epro software

INTERVENTIONS:
Device: Epro software — EPRO software：patients with symptoms will fill in report forms via the software, when the data upload to the terminal, the doctor according to the results of the upload ePRO corresponding medical assessment,and give advises.
  Arms: Group B

SUMMARY:
After receiving chemotherapy, targeted therapy, immunotherapy and other drug treatments, tumor patients often experience various adverse reactions such as bone marrow suppression, diarrhea, pneumonia, etc. However, due to the limited capacity of the hospital, if patients who are discharged home cannot timely detect and deal with severe drug adverse reactions, it will cause harm to their bodies and even threaten their life safety. With the rapid development of network communication, many foreign institutions have tried to develop ePRO software based on patient symptom reports. This type of software is used to monitor drug adverse reactions and provide timely feedback to the attending physician for medical intervention. Existing studies have shown that the application of this type of ePRO software significantly reduces the severity of drug adverse reactions on patients and significantly prolongs survival time.

In this study, the investigators plan to collaborate with Shenzhen 123 Digital Medical Group Co., Ltd. to design and develop a tumor ePRO software that allows outpatient treatment period patients who are discharged home to regularly self-assess the severity of drug adverse reactions and automatically feed back the scoring results to the department's monitoring center. Doctors will make timely diagnosis and treatment based on each patient's score results in order to maximize patient safety after treatment at home. The results of this study will provide better follow-up care for tumor patients who are discharged home after anti-tumor treatment by significantly improving the safety of outpatient treatment period patients with tumors and thereby improving patient survival time and quality.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology confirmed as malignant tumor;
2. ECOG (Eastern Cooperative Oncology Group) performance status score: 0-1;
3. The expected survival time was ≥6 months;
4. Intended to receive systemic antitumor therapy (Cisplatin/oxaliplatin regimen);
5. Proficient in using ePRO software after training;

Exclusion Criteria:

1. Patients who were unable to operate the ePRO system without compliance or after repeated training
2. The chemotherapy regimen did not contain cisplatin or oxaliplatin
3. According to the investigator's assessment, the subjects had other factors that might lead to their forced termination of the study, such as non-compliance with the protocol, other serious diseases requiring combined treatment, serious abnormal laboratory test values of clinical significance, family or social factors, and circumstances that may affect the safety of the subjects or the collection of trial data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Change of health-related quality of life | 3 weeks after taking part in this clinical trial
  Use EThe EORTC QLG Core Questionnaire（EORTC QLQ-C30 ）to evaluate the effect of ePRO software on the quality of life of patients during the chemotherapy period.
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients.The scale contains 30 questions, including treatment response, physical symptoms, mental state, etc. The first 28 options were scored on a scale of 1-4, with a low score indicating a good quality of life or mild symptoms; The last two questions is about Quality of life or health which were scored on a scale of 1-7, with lower scores indicating poorer quality of life or health.

SECONDARY OUTCOMES:
Compliance | 3 weeks after taking part in this clinical trial
  To evaluate the compliance of ePRO software in patients during clinical trial.During this clinical trial the investigators will offer the same electronic questionnaire to both two groups.At the end of the study, the researchers will analyze the proportion of patients in the two groups who completed the questionnaire.A higher percentage of completions in that group means better compliance
Incidence of treatment-related severe adverse reactions | 3 weeks after taking part in this clinical trial
  The effect of ePRO software on the incidence of treatment-related severe adverse reactions.At the end of the study, the researchers will compare the adverse reactions that occurred during the trial between the two groups of patients according to ctcae4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shikai Wu, Principal Investigator — Peking Univerisity First Hospital
Locations (1):
- Peking University First Hospital Ethics Committee, Beijing, Beijing Municipality, China